CLINICAL TRIAL: NCT05770804
Title: The Effect of Education Given to Young Women on Sexual and Reproductive Health Knowledge and Stigma Levels: A Randomized Controlled Study
Brief Title: Young Women on Sexual and Reproductive Health Knowledge and Stigma Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Metin Yildiz, Nurse (Asst.Prof.Dr.), Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SakaryaU-metinyildiz-004
Record Dates: First submitted 2023-02-02; First posted 2023-03-15 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Sexuality; Stigmatization; Inflammation
Keywords: sexual health; knowledge; Stigma
MeSH Terms: conditions — Sexuality; Stereotyping; Inflammation; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Face to face group
  Interventions: Behavioral: Face to face education
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Face to face education — Face-to-face training was provided and supported by booklets.
  Arms: Intervention group

SUMMARY:
Aim: Failure to exercise reproductive and sexual rights can increase the risk of unwanted pregnancies, HIV and sexually transmitted infections, sexual coercion and violence, especially in young women. All of these situations affect the physical and mental health of young girls, as well as the health of their families.For this reason, The Effect of Education Given to Young Women on Sexual and Reproductive Health Knowledge and Stigma Levels: A Randomized Controlled Study was planned.

Material and method: The research was conducted as a randomized controlled experimental study. The universe of the research consisted of female students studying at the Faculty of Health Sciences of Ağrı İbrahim Çeçen University between January and June 2022. The sample consisted of individuals who were studying at the Faculty of Health Sciences of Ağrı İbrahim Çeçen University between the same dates and who met the inclusion criteria of the research. "Descriptive Feature Form", "Sexual and Reproductive Health Stigma Scale for Young Women" and sexual health knowledge test were used to collect data. In the analysis of data; percentile distribution, chi-square, Fisher-Freeman- Halton Exact test, paired samples test, t-test in independent groups, Friedman Test, One Way ANOVA test, and post hoc analyzes (Bonferroni, Games Howell, Dunn) were used.

ELIGIBILITY:
Inclusion Criteria: Be between the ages of 18-24. Agree to participate voluntarily. -

Exclusion Criteria: be over 24 years old

-

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Face to face group | 6 weeks
  2. The Stigma of Sexual and Reproductive Health in Young Women Scale (SCASS): Hall et al. It was developed by in 2017 to identify the stigma of sexual and reproductive health in women aged 15-24. The original scale consists of 20 items and three sub-dimensions: Accepted stigma, Internalized Stigma, and Attitudes on which Stigma is Based. The accepted stigma sub-dimension consists of a total of 6 items. The lowest score that can be obtained from this dimension is 0, and the highest score is 7. The lowest score that can be obtained from the total of the scale is 0, and the highest score is 20. Each item of the scale is rated as 0=Disagree, 0=Neutral, 1=Agree. The higher the score, the higher the level of stigmatization. An increase in the score obtained from the scale indicates an increase in stigma. The Cronbach alpha value of the scale is 0.74. It is stated that the scale is suitable for all social classes.
Face to face group | 6 weeks
  3. Sexual health knowledge test: It was developed by Petili and Gölbaşı in 2017, and its validity-reliability has been made. The test consists of 40 multiple-choice questions and includes 12 sub-dimensions. During the implementation of the CSBT, the participants are asked to carefully read each question and mark the answer they think is correct. Each answer marked correctly by the participant is scored as "1", and each answer marked incorrectly or left blank is scored as "0". The lowest score that can be obtained from CSBT is 0, and the highest score is 40. It is accepted that the higher the score, the higher the level of sexual health knowledge. The Cronbach alpha reliability coefficient of the test was found to be 0.88, and the internal consistency of the test was reported to be high reliability (Evcili & Gölbaşı, 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Metin YILDIZ, Asst.Prof.Dr., Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided